CLINICAL TRIAL: NCT01408706
Title: The Prostate Immobilization Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Taylor (Other)
Responsible Party: Sponsor-Investigator, James Taylor, James Taylor, MD, Wheaton Franciscan Healthcare
Organization: Wheaton Franciscan Healthcare (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-019-ASH
Record Dates: First submitted 2011-07-25; First posted 2011-08-03 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Adenocarcinoma of the Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miller enema air tip (Active Comparator): The Miller enema air tip rectal balloon is inserted into the rectum prior to radiation simulation and also prior to each radiation treatment to immobilize prostate gland and displace rectal tissue during radiation therapy.
  Interventions: Device: Miller Air tip
- Radiadyne Immobilizer (Active Comparator): The Radiadyne Immobilizer Treatment Device is inserted into the rectum prior to radiation simulation and also prior to each radiation treatment to immobilize prostate gland and displace rectal tissue during radiation therapy
  Interventions: Device: Radiadyne Immobilizer

INTERVENTIONS:
Device: Miller Air tip — Miller Enema Air Tip is inserted into rectum prior to simulation and each radiation treatment.
  Other Names: Miller Enema Air Tip
  Arms: Miller enema air tip
Device: Radiadyne Immobilizer — Radiadyne Immobilizer is inserted into rectum prior to simulation and each radiation treatment
  Arms: Radiadyne Immobilizer

SUMMARY:
The purpose of this study is to compare reproducibility of the device position and location of the prostate rectum interface between two immobilization devices for radiation therapy of prostate carcinoma.

DETAILED DESCRIPTION:
The investigator assessed the device position and location of the interface between rectum and prostate weekly during the course of treatment. This information was obtained using a conebeam CT scan on the treatment couch prior to a regularly scheduled radiation treatment. The conebeam CT scan is a standard tool for monitoring patient position and radiation treatment accuracy. Prior to each radiation treatment, the patient was placed in a vaclock immobilization device, then aligned with room lasers to skin tattoos. On board portal imaging was then employed using the KvKv match technique to place isocenter as simulated. For intact prostate treatment, alignment was made to implanted gold fiducial markers. For post prostatectomy patients, the alignment was to pelvic bony anatomy. After patient alignment was complete, a conebeam CT scan was obtained. The position of the anterior rectal wall and the interface between prostate and rectum was compared to the position of these structures at the time of simulation. Measurement was taken in the midline of the prostate gland between its base and apex of the maximum deviation of the rectum prostate interface from its position at the time of simulation. For post prostatectomy patients, a measurement was taken of the maximum deviation from simulation of interface between the rectum and the prostate bed/bladder. These measurements were recorded weekly by the treating radiation oncologist on the Physician Data Sheet.

The difficulty of device insertion, positioning and inflation was recorded daily by the treating personnel based on a scale in the PIDS Daily Radiation Therapist Questionnaire, from 1(none) to 5(unable to insert). These results were summarized by the clinical study coordinators on the PIDS Radiation Therapist Summary.

Patient expression of discomfort during device placement was recorded daily by treating personnel based on a scale in the PIDS Daily Radiation Therapist Questionnaire, from 1(none) to 5(intolerable). These responses will be summarized by the clinical study coordinators on the PIDS Radiation Therapist Summary.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinically localized T1-3 N0-1 M0 adenocarcinoma of the prostate
* Planned definitive radiation therapy

Exclusion Criteria:

* Prior proctectomy
* Rectal surgery within one year
* Proctitis
* Rectal carcinoma
* Anal Stenosis
* History of inflammatory bowel disease
* Scleroderma
* Systemic sclerosis
* Refusal of treatment with immobilization device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Taylor, MD, Principal Investigator — Wheaton Franciscan Cancer Care - All Saints
Locations (1):
- Wheaton Francsican Cancer Care - All Saints, Racine, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Miller Enema Air Tip: Use of Miller enema air tip to fix prostate location and displace rectal tissue during radiation therapy.
  Prostate gland immobilization with rectal balloon: Device: Prostate gland immobilization with rectal balloon (Miller enema air tip or Radiadyne Prostate Immobilizer Treatment Device) to fix prostate location and displace rectal tissue during radiation therapy.
- Radiadyne Immobilizer Treatment Device: Use of Radiadyne Immobilizer Treatment Device to fix prostate location and displace rectal tissue during radiation therapy
  Prostate gland immobilization with rectal balloon: Device: Prostate gland immobilization with rectal balloon (Miller enema air tip or Radiadyne Prostate Immobilizer Treatment Device) to fix prostate location and displace rectal tissue during radiation therapy.
Period: Overall Study
Arm/Group | Miller Enema Air Tip | Radiadyne Immobilizer Treatment Device
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miller Enema Air Tip | Radiadyne Immobilizer Treatment Device | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 23 | 23 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Clinically localized T1-3, NO, MO adenocarcinoma of the prostate [Number; unit: participants] | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Deviation of the Prostate Rectal Interface From Its Position at Time of Simulation.
Description: Measurements will be taken for at least 5, and up to 9, occasions on a weekly basis during each patient's course of treatment. An average value will be determined for each patient. An average of individual patient values will be determined for each immobilization device.
Time Frame: Up to 9 weeks
Measure: Mean (Standard Deviation); unit: CENTIMETERS
Arm/Group | Miller Enema Air Tip | Radiadyne Immobilizer Treatment Device
Number analyzed (Participants) | 29 | 30
CENTIMETERS | .319 (.603) | .095 (.202)

2. Secondary Outcome: Difficulty of Insertion.
Description: Difficulty of device insertion was scored for each treatment by the treating radiation therapist on a scale from 1(easiest) to 5(most difficult). An average score was obtained at completion of therapy for each patient. At completion of the study, an average value was obtained for each immobilization device by averaging the average score for each patient .
Time Frame: Up to nine weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Miller Enema Air Tip | Radiadyne Immobilizer Treatment Device
Number analyzed (Participants) | 29 | 30
units on a scale | 1.083808 [1 to 5] | 1.067535 [1 to 5]

3. Secondary Outcome: Patient Expression of Discomfort
Description: Patient expression of discomfort was scored for each insertion by the treating radiation therapist on a scale from 1(none) to 5(intolerable). An average score was obtained at completion of therapy for each patient. At completion of the study, an average value was obtained for each immobilization device by averaging the average score for each patient .
Time Frame: Up to nine weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Radiadyne Immobilizer Treatment Device: The Radiadyne Immobilizer Treatment Device is inserted into the rectum prior to radiation simulation and also prior to each radiation treatment to immobilize prostate gland and displace rectal tissue during radiation therapy
Arm/Group | Miller Enema Air Tip | Radiadyne Immobilizer Treatment Device
Number analyzed (Participants) | 29 | 30
units on a scale | 1.138237 [1 to 3] | 1.087719 [1 to 3]

ADVERSE EVENTS:
Time Frame: up to nine weeks
Description: Investigator interviews patient weekly during treatment with exam as needed to assess for adverse events.
Arm/Group | Miller Enema Air Tip | Radiadyne Immobilizer Treatment Device
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No